CLINICAL TRIAL: NCT01277731
Title: Pilot Study of Methylprednisolone Replacement for Dexamethasone-induced Hiuup Patients
Brief Title: Methylprednisolone Replacement for Dexamethasone-induced Hiccup
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hun Kang, Associate Professor, Gyeongsang National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gyeongsang-20100701
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Dexamethasone; Hiccup
MeSH Terms: conditions — Hiccup | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylprednisolone replacement (Experimental): This study will enroll the patients who were previously experienced dexamethasone-induced hiccup. Patients who experienced dexamethasone-induced hiccup during chemotherapy will enroll to study arm.
  Run-in period * Dexamethasone 10mg-20mg q day iv during chemotherapy
  ▶ measure hiccup and nausea/vomiting severity
  Treatment period * Methylprednisolone 60mg-125mg iv during chemotherapy
  ▶ measure hiccup and nausea/vomiting severity
  Response will be evaluated by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) and NRS to hiccup at 24hrs after start methylprednisolone.
  Nausea and vomiting will be assessed as CTCAE 4.0
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Run-in period: dexamethasone 10-20mg q day iv during chemotherapy Treatment period: methylprednisolone 60-125mg iv during chemotherapy

SUMMARY:
Dexamethasone is a potent synthetic member of the corticosteroid. It is given to cancer patients undergoing chemotherapy to counteract emetic side effect and essential drug for the chemotherapy-treated patients. Hiccup is common adverse effect of corticosteroid especially on dexamethasone varying from 3% to 60% of given patients. Discontinuance of dexamethasone relieves most hiccupping cases, but vomiting/nausea rates increase. It is not clear whether hiccup side effect is limited to the dexamethasone only or other corticosteroid group.

Methylprednisolone, synthetic corticosteroid as similar as dexamethasone, could be considered as antiemetic agent for the patients with receiving chemotherapy. The investigators perform this pilot study under hypothesis that replacing dexamethasone with methylprednisolone could maintain antiemetic role and prevent hiccup.

ELIGIBILITY:
Inclusion Criteria:

* Age olderthan 21
* A Patient on chemotherapy who was diagnosed malignant tumor
* A Patient who is newly developed hiccup in the course of chemotherapy
* A patient with the willingness to comply with the study protocol during the study period and capable of ccomplying with it
* A patient who signed the imformed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages

Exclusion Criteria:

* A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications
* A patient with uncontrolled diabetes
* A patient who developed uncontrolled serious infection or other uncontrolled serious concomitant diseases
* A patient with disease progression after run-in period who is expected to receive another chomotherapeutic agents with different level of emetic risk

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Prevention rate of dexamethasone induced hiccup | 24hrs after chemotherapy
  measure the presence of hiccup and its severity 24 hous after chemotherapy

SECONDARY OUTCOMES:
Prevention rate of nausea and vomiting | acute; 24 hours, delayed; 7 days after chemotherapy
  Prevention rate of nausea and vomiting 24 hours and 7 days after chemotherapy, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hun Kang, M.D, Ph.D, Principal Investigator — Gyeongsang University Hospital
Locations (1):
- Gyeongsang University Hospital, Jinju, South Korea